CLINICAL TRIAL: NCT02537717
Title: A Contralateral Dispensing Clinical Trial of Study Test Silicone Hydrogel Lens Against Enfilcon A Silicone Hydrogel Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV-15-55
Record Dates: First submitted 2015-08-27; First posted 2015-09-02 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sapphire lens (Experimental): Each subject will be randomized to wear the test lens in one eye and control lens in the other eye. Both test and control lenses will be used in a daily wear modality for one month.
  Interventions: Device: Sapphire Lens
- enfilcon A (Active Comparator): Each subject will be randomized to wear the test lens in one eye and control lens in the other eye. Both test and control lenses will be used in a daily wear modality for one month.
  Interventions: Device: enfilcon A

INTERVENTIONS:
Device: Sapphire Lens — Each subject randomized to wear either the test or control in either the left of right eye.
  Arms: Sapphire lens
Device: enfilcon A — Each subject randomized to wear either the test or control in either the left of right eye.
  Arms: enfilcon A

SUMMARY:
This will be a 1-month dispensing, double-masked, randomized, contralateral study comparing the test lens against the control lens. The assignment of lenses to eyes (i.e. which lens type is to be worn in which eye throughout the study) will be selected according to a randomization table.

DETAILED DESCRIPTION:
Both test and control lenses will be used in a daily wear modality for 1 month. It is anticipated that this study will involve the following visits: Baseline (screening and dispense visit combined), 2-week visit and 4-week visit.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age and has full legal capacity to volunteer
* Has read and understood the information consent letter
* Is willing and able to follow instructions and maintain the appointment schedule
* Is correctable to a visual acuity of 20/30 or better (in each eye) with their habitual correction or the assigned study lenses
* Is an adapted soft contact lens wearer (For the purpose of this study: Current lens wear at least 3 days per week, 8 hours each day.)

Exclusion Criteria:

* Is participating in any concurrent clinical or research study
* Has any known active* ocular disease and/or infection;
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable
* Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable^
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study
* Is pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit). Rationale is that systemic changes over time due to pregnancy/lactating may adversely affect contact lens wear e.g. ocular dryness may increase.
* Is aphakic
* Has undergone corneal refractive surgery.

For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Participants will be excluded with significant slit lamp findings (e.g. infiltrates or other slit lamp findings Grade 3 or above: corneal edema, tarsal abnormalities, and conjunctival injection) or active ocular disease (e.g. glaucoma, history of recurrent corneal erosions, and intraocular infection or inflammation of an allergic, bacterial, or viral etiology).

^ For the purposes of this study, participants will be excluded, if currently taking medication, such as oral antihistamines, antihistamine eye drops, oral and ophthalmic beta-adrenergic blockers (e.g. Propanolol, Timolol), anticholinergics, oral steroids and any prescribed or over-the-counter eye medication, except artificial tears or eye lubricants

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, Principal Investigator — University of Waterloo
Locations (1):
- Center for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Each subject will be randomized to wear the test lens in one eye and control lens in the other eye. Both test and control lenses will be used in a daily wear modality for one month.
  Sapphire Lens: Contact lens. Enfilcon A: contact lens
Period: Overall Study
Arm/Group | Overall Study
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 17

OUTCOME MEASURES:

1. Primary Outcome: Subjective Ratings of Comfort
Description: Subjective ratings of Comfort on a scale (0-100) assessed : 0= Cannot be worn, causes pain, 20=Frequently irritating, 40= Occasionally irritating, 60= Occasionally noticable but not irritating, 80= rarely noticeable, 100= cannot be felt ever
Time Frame: Baseline (After 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- Sapphire Lens: Each subject will be randomized to wear the test lens in one eye and control lens in the other eye. Both test and control lenses will be used in a daily wear modality for one month.
  Sapphire Lens: Contact lens
- Enfilcon A: Each subject will be randomized to wear the test lens in one eye and control lens in the other eye. Both test and control lenses will be used in a daily wear modality for one month.
  enfilcon A: contact lens
Arm/Group | Sapphire Lens | Enfilcon A
Number analyzed (Participants) | 17 | 17
Number analyzed (eyes) | 17 | 17
units on a scale | 92 (9) | 91 (9)

2. Primary Outcome: Subjective Ratings of Comfort
Description: as for outcome 1
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Sapphire Lens | Enfilcon A
Number analyzed (Participants) | 17 | 17
Number analyzed (eyes) | 17 | 17
units on a scale | 80 (18) | 82 (8)

3. Primary Outcome: Subjective Ratings of Comfort
Description: as for outcome 1
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Sapphire Lens | Enfilcon A
Number analyzed (Participants) | 17 | 17
Number analyzed (eyes) | 17 | 17
units on a scale | 81 (16) | 80 (14)

4. Primary Outcome: Subjective Comfort Preference
Description: Subjective comfort preference Sapphire lens, Enfilcon A, no preference
Time Frame: Baseline (after 10 minutes of lens dispense)
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Overall Study
Number analyzed (Participants) | 17
Number analyzed (Eyes) | 34
percentage of eyes
  Sapphire lens | 47
  enfilcon A | 12
  No preference | 41

5. Primary Outcome: Subjective Comfort Preference
Description: Subjective comfort preference Sapphire lens, Enfilcon A, no preference
Time Frame: 2 weeks
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Overall Study
Number analyzed (Participants) | 17
Number analyzed (Eyes) | 34
percentage of eyes
  Sapphire lens | 53
  enfilcon A | 18
  No preference | 29

6. Primary Outcome: Subjective Comfort Preference
Description: Subjective comfort preference Sapphire lens, Enfilcon A, no preference
Time Frame: 4 weeks
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Overall Study
Number analyzed (Participants) | 17
Number analyzed (Eyes) | 34
percentage of eyes
  Sapphire lens | 47
  enfilcon A | 18
  No preference | 35

7. Primary Outcome: Lens Wettability
Description: Lens wettability was assessed on a Grading scale (0-4, 0.25 steps) (0=excellent; 4=severely reduced)
Time Frame: Baseline (After 10 minutes of lens dispense)
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Sapphire Lens | Enfilcon A
Number analyzed (Participants) | 17 | 17
Number analyzed (eyes) | 17 | 17
units on a scale | 2.9 (0.7) | 2.6 (1.0)

8. Primary Outcome: Lens Wettability
Description: Lens wettability was assessed on a Grading scale (0-4, 0.25 steps) (0=excellent; 4=severely reduced)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Sapphire Lens | Enfilcon A
Number analyzed (Participants) | 17 | 17
Number analyzed (eyes) | 17 | 17
units on a scale | 2.8 (1.0) | 2.8 (0.8)

9. Primary Outcome: Lens Wettability
Description: Lens wettability was assessed on a Grading scale (0-4, 0.25 steps) (0=excellent; 4=severely reduced)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Sapphire Lens | Enfilcon A
Number analyzed (Participants) | 17 | 17
Number analyzed (eyes) | 17 | 17
units on a scale | 2.9 (0.9) | 2.6 (1.0)

ADVERSE EVENTS:
Time Frame: From dispense up to one month on study lenses
Arm/Group | Sapphire Lens | Enfilcon A
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No